CLINICAL TRIAL: NCT04184375
Title: Evaluation of Cognitive Stimulation on Dysexecutive Residual Symptoms in Bipolar Patients Over 65 Years of Age
Brief Title: Cognitive Stimulation for Elderly Bipolar Patients
Acronym: TONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015/P05/095
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Disorder; Cognitive Impairment; Age-related Cognitive Decline
MeSH Terms: conditions — Bipolar Disorder; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TONIC (Experimental): The cognitive stimulation sessions are carried out using Liliane Israël's "TRAIN YOUR MEMORY" software, and are divided into two parts: the first part is essentially cognitive and the second relates to the daily life of the Bipolar patient.
  This training method consists of combining two means of intervention, pedagogical action and psychotherapeutic effect. It aims to stimulate, develop and strengthen the basic mechanisms underlying memory phenomena (sensory acuity, attention, associations, structuring, executive functions, spatial and temporal landmarks, associative recruitment). It is presented in the form of exercises divided into eight modules.
  Interventions: Behavioral: cognitive stimulation
- Control (No Intervention): The usual practice consists of interviews with the psychiatrist with the possibility of home visits by the nurse.

INTERVENTIONS:
Behavioral: cognitive stimulation — Patients participate in one session per week according to the following schedule:
  * 2 sensory stimulation sessions: identify sensations, emotions, how to manage them.
  * 2 sessions on association, verbal fluency, and imagination: language as a tool for expression in the face of illness.
  * 2 voluntary attention sessions: improve daily attention.
  * 2 sessions of intellectual structuring: stimulating and maintaining memory, carrying out external activities.
  * 2 sessions of structuring through language: impact on social life.
  * 2 sessions stimulating the temporal and spatial landmarks: agenda, daily trips.
  Arms: TONIC

SUMMARY:
Age is a major risk factor for the development of cognitive disorders and neurodegenerative pathologies. Cognitive disorders during the phases of bipolar disease are known to exist, and alterations increase significantly after the age of 65. Drug treatments seem to have only a limited effect. A cognitive stimulation program has proven his benefit to patients over 65 with neurodegenerative diseases (Israel, 2004). We propose to evaluate this cognitive stimulation program that we have adapted to bipolar disease.

DETAILED DESCRIPTION:
Bipolar disorders, which belong to the category of mood disorders, are the 6th leading cause of disability in the world. Cognitive disorders are known to exist during the phases of bipolar disease, and alterations increase significantly after the age of 65. Recent studies have shown that attention, memory and executive function impairments are the main causes of cognitive disorders. Residual symptoms have a significant impact on the risk of relapse into bipolar disorder and on quality of life. Cognitive stimulation (CS) is a pedagogical approach based on the idea that cognitive skills contribute to personal development in the same way as psychological and social factors. This study aims at assessing a cognitive stimulation program initially developed for patients with neurodegenerative diseases, and adapted to bipolar disease. This program will be compared to the usual practice consisting in consultation with psychiatrist and sometimes in intervention of home nurses.

ELIGIBILITY:
Pre-Inclusion Criteria:

* age > 65 years old
* Diagnosis of bipolar illness for more than 10 years
* Euthymic phase
* Understands and speaks French
* Free, informed and express consent

Inclusion Criteria:

* Mild to moderate neuro-cognitive impairments (MMS Test : 16 ≤ score < 26)

Exclusion Criteria:

* Illiteracy
* Patient participating in other therapeutic workshops (e. g. psycho-geriatric day hospital care, etc.)
* Persons deprived of their liberty by a judicial or administrative decision
* Persons of full age who are subject to a legal protection measure
* Persons unable to consent
* Persons who are not members of or beneficiaries of a social security scheme
* Patient's refusal to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
Score at the Frontal Assessment Battery (FAB) | at 3 months after inclusion
  The FAB assesses conceptualization (category responses, such as "in what way are a banana and an orange are alike?"), lexical fluency, programming or motor series (Luria), sensitivity to interference (conflicting instructions, such as "tap twice when I tap once"), inhibitory control (Go/No-Go), and environmental autonomy (prehension behavior, such as "do not take my hands")

SECONDARY OUTCOMES:
Score at FAB | at 6 months after inclusion
  Scores between the 3-month and 6-month evaluation will determine whether executive analysis functions have been maintained
Number of patients with a positive difference between the scores on the Functional Activities Questionnaire (QAF) | at inclusion
  The QAF allows to quickly assess a patient's functional capacity and to identify a functional decline in the patient with a mild neurocognitive disorder, Alzheimer's disease or other neurocognitive disorder.
Number of patients with a positive difference between the scores on the Functional Activities Questionnaire (QAF) | at 6 months after inclusion
  A positive difference in scores reflects an improvement in patient autonomy
Score at delayed matching-to-sample (DMS48) | at inclusion
  The DMS48 is a test of visual recognition memory test
Score at DMS48 | at 3 months after inclusion
  The DMS48 is a test of visual recognition memory test
Time in minutes at the Trail Making Test A (TMTA) | at inclusion
  Evaluation of speed of processing.
Time in minutes at the Trail Making Test A | at 3 months after inclusion
  Evaluation of speed of processing.
Number of errors at Trail Making Test B (TMTB) | at inclusion
  Evaluation of mental flexibility
Number of errors at Trail Making Test B (TMTB) | at 3 months after inclusion
  Evaluation of mental flexibility
Score at ISAAC test | at inclusion
  Measures fluence
Score at ISAAC test | at 3 months after inclusion
  Measures fluence
Score at Montreal Cognitive Assessment (MMS) | at inclusion
  Assessment for detecting cognitive impairment
Score at Montreal Cognitive Assessment (MMS) | at 6 months after inclusion
  Assessment for detecting cognitive impairment
Score at the Hamilton Depression Rating Scale | at inclusion
  Evaluation of patient thymic state
Score at the Hamilton Depression Rating Scale | at 6 months after inclusion
  Evaluation of patient thymic state
Interference score at the Stroop test | at inclusion
  Evaluation of selective attention
Interference score at the Stroop test | at 6 months after inclusion
  Evaluation of selective attention
Number of hospitalization due to relapse | at 6 months after inclusion
  hospitalization due to relapse
Score at Zarit scale (caregiver) | at inclusion
  Identification of suffering or exhaustion, anxiety and/or depressive disorder(s), sleep disorder(s), etc. in the caregiver
Score at Zarit scale (caregiver) | at 6 months after inclusion
  Identification of suffering or exhaustion, anxiety and/or depressive disorder(s), sleep disorder(s), etc. in the caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Puzos, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (1):
- Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available with publication. A Digital Object Identifier will be used.
  Keyword are bipolar disorder, aged, cognitive dysfunction, cognitive Remediation.
  The only available version will be the locked database. With the exception of dates, all data will be made available. Dates will only be collected to verify the quality of the clinical trial execution. They do not add to the clinical question, and may be a means of indirectly identifying patients. The database will be made available through Mendeley Data.
  Medical Subject Headings (MESH) terms will be used to describe clinical data. Psychological test references will be provided in the publication. International standard unit will be used. The data will be made available to the community of scientists and clinicians interested in bipolar disorder.
  Data will be made available with the free access to the publication for 15 years.
Supporting Information: CSR
Time Frame: Data will be made available with publication and up to 15 years after the end of the study
Access Criteria: On Mendeley repository A Digital Object Identifier will be provided